CLINICAL TRIAL: NCT05654870
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Valbenazine as Adjunctive Treatment in Subjects With Schizophrenia
Brief Title: Study to Evaluate the Efficacy, Safety, and Tolerability of Valbenazine as an Adjunctive Treatment for Schizophrenia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study ATS3020 was closed due to business reasons. Neurocrine Biosciences will continue to conduct study ATS3019 (NCT05110157). There were no unexpected safety findings for this compound that motivated the decision.
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBI-98854-ATS3020
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Schizophrenia
Keywords: schizophrenia; valbenazine; antipsychotic; VMAT2; NBI-98854; dopamine; PANSS; Adjunctive
MeSH Terms: conditions — Schizophrenia | interventions — valbenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Valbenazine (Experimental): Valbenazine once daily
  Interventions: Drug: Valbenazine
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valbenazine — Oral treatment
  Other Names: NBI-98854
  Arms: Valbenazine
Drug: Placebo — Placebo matching valbenazine
  Arms: Placebo

SUMMARY:
This primary objective for this study is to evaluate the effect of adjunctive valbenazine versus placebo on symptoms of schizophrenia in participants who have inadequate response to antipsychotic treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Medically confirmed diagnosis of schizophrenia
* Participant is receiving a stable regimen of background antipsychotic medication
* Plasma levels for at least 1 of the participant's antipsychotic medications must be detectable by an available assay
* Participant is an outpatient with stable symptomatology
* Participant must have an adult informant (for example, a family member, relative, partner, social worker, caseworker, residential facility staff, or nurse)

Key Exclusion Criteria:

* Has a history of treatment resistant schizophrenia
* Have a clinically significant unstable medical condition in the judgement of the investigator or any laboratory value outside the normal range that is considered by the investigator to be clinically significant at the screening visit
* Prior (within 6 months of Screening) or concomitant use of any vesicular monoamine transporter 2 (VMAT2) inhibitor (that is, valbenazine, reserpine, tetrabenazine, deutetrabenazine); or a history of intolerance to VMAT2 inhibitors

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Change in Positive and Negative Syndrome Scale (PANSS) Total Score from Baseline to Week 10 | Baseline, Week 10

SECONDARY OUTCOMES:
Change in Clinical Global Impression of Severity (CGI-S) Score from Baseline to Week 10 | Baseline, Week 10
Change in Personal and Social Performance (PSP) Score from Baseline to Week 10 | Baseline, Week 10

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (3):
- United States (3):
  - Neurocrine Clinical Site, San Jose, California
  - Neurocrine Clinical Site, Coral Gables, Florida
  - Neurocrine Clinical Site, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No